CLINICAL TRIAL: NCT06230809
Title: Internet Based Self-help for Problem Gambling Concerned Significant Others
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The National Gambling Helpline Sweden (Unknown)
Responsible Party: Principal Investigator, Anders Nilsson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-04225-01
Record Dates: First submitted 2023-10-02; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Problem Gambling
Keywords: concerned significant others

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Web-based self-help
- Waitlist (No Intervention): Waitlist, participants will be included after 8 weeks.

INTERVENTIONS:
Behavioral: Web-based self-help — Web-based self-help with 5 modules, lasting 5 weeks.
  Arms: Intervention

SUMMARY:
The project aims to evaluate a brief online self-help intervention for Concerned Significant Others of individuals with Problem Gambling. The intervention consists of five modules with texts, films and exercises and is compared to a waiting list.

ELIGIBILITY:
Inclusion Criteria:

* No treatment related to the gambling during the past 3 months for the CSO
* The CSO is at least 18 years old
* The CSO can read and answer questions in Swedish.
* The CSO is assessed as a non-problem gambler according to the Gambling Disorder Identification Test.

Exclusion Criteria:

* Displaying symptoms of severe psychiatric disorders such as psychosis or bipolar disease deemed to needed other treatment options.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Kessler-9 | At baseline and post treatment (5-7 weeks after inclusion) and again 3, 6, and 12 months following treatment completion
  Mental health

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | At baseline and post treatment (5-7 weeks after baseline) and again 3, 6, and 12 months following treatment completion
  Depressive symptoms
Generalized Anxiety Disorder 7-item scale | At baseline and post treatment (5-7 weeks after inclusion), and again 3, 6, and 12 months following treatment completion
  Anxiety symptoms
Relationship Assessment Scale | At baseline and post treatment (5-7 weeks after inclusion), and again 3, 6, and 12 months following treatment completion
  Relationship satisfaction
Family Member Impact Scale | At baseline and post treatment (5-7 weeks after inclusion), and again 3, 6, and 12 months following treatment completion
  Gambling-related family stress
Coping Questionnaire | At baseline and post treatment (5-7 weeks after inclusion), and again 3, 6, and 12 months following treatment completion
  Coping
Brunnsviken Brief Quality of life quality scale | At baseline and post treatment (5-7 weeks after inclusion), and again 3, 6, and 12 months following treatment completion
  Quality of life

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request.